CLINICAL TRIAL: NCT02805231
Title: Associations of Vitamin D Receptor Polymorphisms With the Risk of Primary Open-angle Glaucoma
Brief Title: Associations of Vitamin D Receptor ApaI and Tru9I Polymorphisms With the Risk of Primary Open-angle Glaucoma
Status: Completed | Type: Observational
Sponsor: Lv Yingjuan (Other)
Collaborators: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Sponsor-Investigator, Lv Yingjuan, department of ophthamology, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Other Study IDs: tjykdxykyy4
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Primary Open- Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — ApaI and Tru9I Polymorphisms

GROUPS / COHORTS (2):
- primary open-angle glaucoma patients: vitamin D receptor polymorphic analysis was studied by real-time polymerase-chain reaction high resolution melting analysis in primary open-angle glaucoma patients.
  Interventions: Other: Vitamin D receptor polymorphic analysis
- randomly age-matched people: vitamin D receptor polymorphic analysis was studied by real-time polymerase-chain reaction high resolution melting analysis in randomly age-matched people.
  Interventions: Other: Vitamin D receptor polymorphic analysis

INTERVENTIONS:
Other: Vitamin D receptor polymorphic analysis

SUMMARY:
This study investigated whether vitamin D receptor gene polymorphism is altered in primary open-angle glaucoma subjects carrying the risk allele.Primary open-angle glaucoma patients and age-matched people in the Han population were enrolled. Vitamin D receptor polymorphic analysis was studied by polymerase chain reaction-restriction fragment length polymorphism technique.

ELIGIBILITY:
Inclusion Criteria:

* intraocular pressure greater than 22 mmHg with two or more medications wide anterior chamber angle glaucomatous optic neuropathy (Glaucomatous optic nerve damage was defined as cup-to-disc ratio higher than 0.7 or focal loss of the nerve fiber layer (notch) associated with a consistent glaucomatous visual field defect) visual field loss consistent with optic nerve damage and visual fields were performed by using standard automated perimetry

Exclusion Criteria:

* the presence of any secondary glaucoma including exfoliation syndrome or a history of ocular trauma high myopia macular degeneration other ocular diseases a known history of systemic diseases and administration of vitamin D3 or other analog

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary open-angle glaucoma patients and randomly age-matched people as controls in the Han population of Tianjin China
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
gene polymorphisms of vitamin D receptor | 1 day visit

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China